CLINICAL TRIAL: NCT05133986
Title: Using Untargeted Metabolomics to Identify Urinary Biomarkers of Onion Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manchester Metropolitan University (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elliot Owen, PhD Student, Manchester Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 34047
Record Dates: First submitted 2021-11-02; First posted 2021-11-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Metabolomics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Onion feeding first, couscous feeding second (Experimental): Participants will report to the laboratory at 8am in a fasted state (water consumption is permitted) and provide a spot baseline urine sample. Participants will then be served a 120g portion of onions (experimental condition), prepared under standardized conditions. Participants shall remain supervised in the laboratory and will only consume water (100mL per hour) for the subsequent 6 hours, after which participants are free to consume their habitual diet (except alcohol, tea coffee, and FVs). In the 24-hour postprandial test period, participants will obtain urine samples at several time-points. Urine collection vessels will be used to obtain samples at 0-1, 1-2, 2-4, 4-6, 6-12, 12-24 hours. This experimental protocol shall be repeated following a 4-day washout period (habitual diet consumption with no restrictions imposed on participants) with 120g of couscous consumed instead of onions, as a control condition.
  Interventions: Other: Onion Feeding; Other: Couscous Feeding
- Couscous feeding first, onion feeding second (Experimental): Participants will report to the laboratory at 8am in a fasted state (water consumption is permitted) and provide a spot baseline urine sample. Participants will then be served a 120g portion of couscous (control condition), prepared under standardized conditions. Participants shall remain supervised in the laboratory and will only consume water (100mL per hour) for the subsequent 6 hours, after which participants are free to consume their habitual diet (except alcohol, tea coffee, and FVs). In the 24-hour postprandial test period, participants will obtain urine samples at several time-points. Urine collection vessels will be used to obtain samples at 0-1, 1-2, 2-4, 4-6, 6-12, 12-24 hours. This experimental protocol shall be repeated following a 4-day washout period (habitual diet consumption with no restrictions imposed on participants) with 120g of onions consumed instead of couscous, as an experimental condition.
  Interventions: Other: Onion Feeding; Other: Couscous Feeding
- Onion supplementation period (Other): This dose-dependent biomarker validation intervention will include three 4-day supplementation periods separated by two 3-day washout periods. Supplementation periods will provide participants with a daily portion of onions to be consumed with their evening meals. The daily quantity of onion supplementation, low (40g), medium, (80g) and high (160g), will remain constant throughout each 4-day period, and the order will be individually randomised. Participants will be asked to avoid onion intake throughout the supplementation periods, other than the portions provided by researchers. First morning void urine samples will be collected by participants on the morning after the supplementation period and obtained by researchers.
  Interventions: Other: Onion Supplementation Period

INTERVENTIONS:
Other: Onion Feeding — The intervention includes feeding individuals a 120g portion of onions (experimental condition).
  Arms: Couscous feeding first, onion feeding second; Onion feeding first, couscous feeding second
Other: Couscous Feeding — The intervention includes feeding individuals a 120g portion of couscous (control condition).
  Arms: Couscous feeding first, onion feeding second; Onion feeding first, couscous feeding second
Other: Onion Supplementation Period — Three 4-day supplementation periods separated by two 3-day washout periods. Supplementation periods will provide participants with a daily portion of onions to be consumed with their evening meals. The daily quantity of onion supplementation, low (40g), medium, (80g) and high (160g), will remain constant throughout each 4-day period, and the order will be individually randomised.
  Arms: Onion supplementation period

SUMMARY:
Fruit and vegetable (FV) intake has been reported as a modifiable risk factor of globally pervasive chronic diseases. Traditionally, the measurement of dietary intake has been conducted via self-report methods such as food diaries, food frequency questionnaires, and dietary recall. These methods are inherently subject to sources of error and biases. The objective measurement of diet-specific urinary biomarkers has been proposed as an alternate assessment method. A dose-dependent biomarker or biomarker panel for total FV intake has been investigated but not successfully established. In a recent publication as part of this PhD research, the researchers outlined a concise panel of 7 FVs that are predictive of total FV intake in a UK population. Recent studies have implemented an untargeted metabolomic approach to identify novel biomarkers of some of the 7 FVs identified in our prior research, but not with onion intake. The aim of this study is to detect, quantify and identify dose-dependent biomarker(s) of onion intake in a UK population using untargeted metabolomics. Phase 1 will be an acute randomised crossover intervention study, involving the consumption of a standardised portion of cooked onions (test) or couscous (control). Urine samples over the 24-hour period post-consumption will be collected. Phase 2 will be a dose-dependent crossover intervention study, where participants are supplied with supplementary onion portions (low, medium, high) to be consumed with their habitual evening meals. Within each supplementation period, participants will consume the same quantity of onions across the 4 days and collect a midstream first void urine samples on the fifth day. Trial order will be randomised, and a washout period of 3 days will be implemented between supplementation periods. 14 participants will be recruited for both phases of data collection. Urine samples will be analysed by high-performance liquid-chromatography with quadrupole time-of-flight mass spectrometry (LC-QTOF-MS) to identify potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-pregnant/lactating
* BMI between 18.5 and 30 kg/m^2
* Non-smokers.

Exclusion Criteria:

* Any diagnosed health condition (chronic or infectious diseases)
* Consumption of medications/nutritional supplements
* Any allergies/intolerances to onions/couscous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Untargeted metabolomics for onion biomarker identification using LC-QTOF-MS. | 24-hours postprandial period following onion or couscous consumption.
  Urine samples will be analysed to putatively identify biomarkers of onion intake by comparison with control samples using high-performance liquid chromatography coupled to a quadrupole time-of-flight mass spectrometer (LC-QTOF-MS). LC-QTOF-MS analysis allows the simultaneous high-resolution measurement of a broad range of metabolites, hence the untargeted nature of the analysis. Multivariate statistical analysis and Partial least squares Discriminant Analysis included in the mass spectrometry software will be used to analyse LC-QTOF-MS results to identify features that best discriminate between test and control conditions.
Dose-dependency and change in concentration of potential biomarkers identified in Primary Outcome 1 | First morning void urine samples following three periods of 4-day onion supplementation.
  First morning void urine samples will be obtained after three separate 4-day periods of supplementing evening meals with 40g, 80g and 160g of onions. The validity of candidate biomarkers from the first phase of the study, Primary Outcome 1, shall be assessed by LC-QTOF-MS - quantifying urinary concentrations following the consumption of multiple doses of onions across a range of servings.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Metropolitan University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owen EJ, Patel S, Flannery O, Dew TP, O'Connor LM. Derivation and Validation of a Total Fruit and Vegetable Intake Prediction Model to Identify Targets for Biomarker Discovery Using the UK National Diet and Nutrition Survey. J Nutr. 2021 Apr 8;151(4):962-969. doi: 10.1093/jn/nxaa406. PMID 33484153